CLINICAL TRIAL: NCT02554500
Title: Effects of Remote Ischemic Preconditioning in Bone Microcirculation
Brief Title: Bone Microcirculation After Remote Ischemic Preconditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Kisch, MD, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-266-5
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Intact Scaphoid Bone; Intact Metacarpal Bone; Fractured Scaphoid Bone; Fractured Metacarpal Bone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Intact scaphoid bone (Experimental): Group A (n=20): Consent-capable male and female patients ≥18 years of age who have an intact scaphoid bone.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
- Intact metacarpal bone (Experimental): Group B (n=20): Consent-capable male and female patients ≥18 years of age who have an intact metacarpal bone.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
- Fractured scaphoid bone (Experimental): Group C (n=20): Consent-capable male and female patients ≥18 years of age who have a fractured scaphoid bone.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
- Fractured metacarpal bone (Experimental): Group D (n=20): Consent-capable male and female patients ≥18 years of age who have a fractured metacarpal bone.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
- Intact metatarsal bone (Experimental): Group B (n=20): Consent-capable male and female patients ≥18 years of age who have an intact metatarsal bone.
  Intervention: Remote Ischemic Preconditioning (by Blood Pressure Cuff)
  Interventions: Procedure: Remote Ischemic Preconditioning (by Blood Pressure Cuff)

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning (by Blood Pressure Cuff) — Remote Ischemik Preconditioning is performed using a Blood Pressure Cuff with a pressure slightly above patients' blood pressure on the upper arm.

SUMMARY:
In trauma surgery and hand surgery treatment strategies of none healing bone fractures aim at replacing pseudarthrosis by well vascularized bone and improving microcirculation. Although previous studies indicate that remote ischemic preconditioning (RIPC) can accelerate bone healing in case of non-union, only a few studies focused on the elucidation of its mechanisms of action. Therefore, the aim of this study is to evaluate the microcirculatory effects of remote ischemic preconditioning (RIPC) on scaphoid bones and metacarpal bones and metatarsal bones in a human in-vivo setting for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Group A (n=20): Consent-capable male and female patients ≥18 years of age who have an intact scaphoid bone.
* Group B (n=20): Consent-capable male and female patients ≥18 years of age who have an intact metacarpal bone.
* Group C (n=20): Consent-capable male and female patients ≥18 years of age who have a fractured scaphoid bone.
* Group D (n=20): Consent-capable male and female patients ≥18 years of age who have a fractured metacarpal bone.

Exclusion Criteria:

* below 18 years of age
* scar tissue above measuring focus
* osteoporosis or comparable bone disease
* medication that influences bones

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Change in microcirculation (composite outcome measure) | Baseline and 1 minute post-dose
  * Bone blood flow [arbitrary units AU]
  * Bone blood velocity [AU]
  * Tissue oxygen saturation [%]
  * Relative postcapillary venous filling pressure [AU] (Composite outcome measure)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany